CLINICAL TRIAL: NCT01788930
Title: Obstructive Sleep Apnea and Aspirin Resistance in Type-2 Diabetic Patients
Brief Title: Aspirin Resistance and Sleep Apnea in Type-2 Diabetic Patients
Acronym: AREAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recommendations changing
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1227
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Atherothrombosis; Type 2 Diabetes; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Thrombosis; Diabetes Mellitus, Type 2; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP (Active Comparator): This device consists in a nasal continuous positive airway pressure (CPAP). It will be applied 3 months after the beginning of drug treatment and for 3 months.
  Other Name: positive airway pressure
  Interventions: Device: CPAP
- Sham-CPAP (Placebo Comparator): This device consists in a sham CPAP. It will be applied 3 months after the beginning of drug treatment and for 3 months.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP

SUMMARY:
Type-2 Diabetes and Sleep Apnea Syndrome (SAS) are both related to an increase in platelet activation. Type 2 diabetes is often associated with sleep apnea syndrome with a prevalence up to 60%.

The main objective of our study is to analyze the influence of sleep apnea on the response to antiplatelet therapy in stable aspirin-treated type-2 diabetes patients.

Consecutive stable aspirin-treated type-2 diabetes patients referred for suspicion of sleep apnea will be recruited after providing informed consent. Response to aspirin will be assessed with the Verify Now Aspirin(TM)rapid analyser in the morning after nocturnal polysomnography, and compared with a group of type-2 diabetes free of sleep apnea. Other endocrine, metabolic, hematologic and cardiovascular confounders will also be assessed at baseline to determine their influence on the response to aspirin.

Then, Patients with severe SAS (Apnea-Hypopnea Index> 30 events/h) and response with Aspirin (ARU > 454) will be randomized to 3 months of active or sham continuous positive airway pressure treatment in a pilot study. After the 3-months of intervention, response to aspirin will be compared between the sham and effective CPAP groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged > 18 years old
* With Type 2 diabetes
* Stable Atherothrombosis for more than 3 months
* Using aspirin for more than 10 days or without aspirin (in this last case, they will do only the observational study.)
* Without any modification in their treatments for 10 days
* Ambulatory patient
* Without any cardiovascular event or inflammatory disease for 3 months before inclusion

Exclusion Criteria:

* Pregnant women
* Other active clinically significant illness, including unstable cardiovascular, or neoplasia which could interfere with the study conduct or counterindicate the study treatments or place the patient at risk during the trial or compromise the study participation
* Patients participating in an other study
* Patient without any medical care insurance
* Any treatment that could interfere with aspirin
* Previous treatment by CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-02; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Response to antiplatelet therapy | Measure will be done in the morning after the sleep diagnosis

SECONDARY OUTCOMES:
Effects of CPAP treatment for severe obstructive sleep apnea on aspirin efficacity in type-2 diabetic patients | Change from baseline after 3 months randomized treatment

CONTACTS AND LOCATIONS:
Overall Officials: Olivier ORMEZZANO, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, Isere, France